CLINICAL TRIAL: NCT01781598
Title: Patient-specific Instruments as a Standard Procedure in Total Knee Arthroplasty: Logistics, Learning Curve, and Postoperative Radiological Results in 70 Patients
Brief Title: Patient-specific Instruments as a Standard Procedure in Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Orthopedic Clinic Gersthof (Other)
Responsible Party: Principal Investigator, Dominik Drnek, Dr. med. univ., Orthopedic Clinic Gersthof
Other Study IDs: PMCBv1
Record Dates: First submitted 2013-01-21; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Alignment
Keywords: Total knee arthroplasty; Patient specific instruments; Patient matched cutting blocks; Alignment; Learning curve; VISIONAIRE
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Patient specific instruments in TKA
  Interventions: Device: Total knee arthroplasty (TKA) (Smith &Nephew®)

INTERVENTIONS:
Device: Total knee arthroplasty (TKA) (Smith &Nephew®)

SUMMARY:
Description of logistics, learning curve and radiological results in 70 patients treated with patient specific instrumentation in total knee arthroplasty as a standard procedure

DETAILED DESCRIPTION:
The Orthopaedic Clinic Gersthof is a teaching hospital, where the entire spectrum of joint replacements with emphasis on hips and knees is performed. Twenty surgeons perform TKAs at our institution, with approximately 400 TKAs implanted per year.

The PSI system of Smith &Nephew® (Patient-Matched Cutting Blocks [PMCB]; the VISIONAIRE® technology) is applied. The preoperative image modality is based on a long leg standing X-ray as well as an MRI of the knee. The Genesis II® Endoprosthesis (Smith & Nephew®) is used as the TKA implant.

This study is a observational monocentric prospective study.

Estimated enrollment: 70 Enrollment time: September 2011-October 2012 Primary outcome: Alignment

The postoperative X-rays (AP, lateral view, and long leg standing), taken 7-to-10 days after surgery are evaluated in terms of component position and restoration of the mechanical alignment. X-rays are routinely monitor-guided but not calibrated at our institution.

As a secondary outcome the learning curve is evaluated using the following parameters collected during surgery: the fit of the cutting blocks, changes of the implant size, bony recuts, soft tissue releases, and changes in inlay size. Gap balancing was subjectively judged by the operating surgeon. Operation time, number of blood transfusions, and early postoperative complications were recorded within the first 14 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Indication for TKA
* Genesis II endoprosthesis
* Operated using patient specific instruments (VISIONAIRE)

Exclusion Criteria:

* contraindication for MRI
* varus/ valgus deformity >15 degrees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with GENESISII prothesis using VISIONAIRE are enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Alignment | Postoperative x-ray (7-10 days after surgery)
  Alignment measured on monitor-guided x-rays:
  Mechanical Alignment: Hip-Knee-Ankle angle in degrees [°] Alignment of the tibial and femoral component in the sagittal and coronal plane [°]

SECONDARY OUTCOMES:
Learning curve | Intraoperative and early postoperative period (up to 14 days after surgery)
  In order to evaluate the learning curve associated with using VISIONAIRE® technology for TKA, the following parameters are registered during surgery: the fit of the cutting blocks[subjective grading by the surgeon], changes of the implant size[number of changes], bony recuts[number of recuts], soft tissue releases[number of releases, kind of release], and changes in inlay size [number of inlay changes]. Gap balancing is subjectively judged by the operating surgeon. Operation time[minutes], number of blood transfusions[units], and early postoperative complications associated with the treatment [kind and number] within the first 14 days after surgery are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Clinic Gersthof, Vienna, Austria